CLINICAL TRIAL: NCT01093638
Title: A Multi-center, Randomized, Double-blinded Clinical Study to Assess the Effect of Insulin Enriched Formula on Gastrointestinal Tract Maturation in Pre-term Infants.
Brief Title: Oral Formulation of Insulin for Preterm Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Elgan Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTILYAB004409LND10LaniadoH
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Premature Birth of Newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Formulation of Insulin (Experimental): Oral formulation of insulin fed concomitantly with premature infant formula
  Interventions: Biological: Oral Formulation of Insulin
- Oral Formulation of Placebo (Placebo Comparator): Oral formulation of placebo fed concomitantly with premature infant formula
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Oral Formulation of Insulin — Oral formulation of insulin fed concomitantly with infant formula
  Arms: Oral Formulation of Insulin
Biological: Placebo — Oral formulation of placebo fed concomitantly with infant formula
  Arms: Oral Formulation of Placebo

SUMMARY:
The study will evaluate the effect of oral formulation of insulin on preterm infants, born between 26-33 weeks of pregnancy, weighing over 750 grams, who meet the inclusion and exclusion criteria established in this protocol.

DETAILED DESCRIPTION:
The study will aim to determine whether an oral formulation of insulin administration enhances gastrointestinal maturation. The gastrointestinal maturation will be evaluated by the ability of premature infants to achieve complete enteral feeds. The insulin concentration administered in the study is physiological and within the insulin concentration range present in human breast milk and colostrum.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-term infants 26-33 weeks gestation.

Ages: 26 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of days to achieve complete enteral feeding | Up to 28 days or discharge and at 3 months of age

SECONDARY OUTCOMES:
Number of gastric residual > 2 ml/kg | Up to 28 days or discharge, at 3 months of age
Number of gastric residual > 50% of previous feeding | Up to 28 days or discharge and at 3 months of age
Number of days to discharge | Up to 28 days or discharge and at 3 months of age
Weight gain | Up to 28 days or discharge and at 3 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Naim Shehadeh, Prof., Study Director — Rambam Health Care Campus
Locations (1):
- NICU, Laniado Hospital, Netanya, Israel

IPD SHARING:
Plan to Share IPD: No